CLINICAL TRIAL: NCT00655096
Title: Screening Protocol for the Evaluation and Diagnosis of Potential Research Participants
Brief Title: Screening for Research Participants
Status: Recruiting | Type: Observational
Sponsor: National Eye Institute (NEI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 080102; 08-EI-0102
Record Dates: First submitted 2008-04-08; First posted 2008-04-09 (Estimated); Last update posted 2025-12-19 (Actual); Status verified 2025-12-12

CONDITIONS: Eye Diseases
Keywords: Eye; Photograph; Retina
MeSH Terms: conditions — Eye Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Affected participants: Adults and children with either diagnosed or un-diagnosed ocular conditions.
- Disease free control: Adults and children without any ocular disorders.
- Unaffected relative: Unaffected first degree relative of a genetic ocular disease participant.

SUMMARY:
This study will allow National Eye Institute (NEI) doctors the opportunity to examine people with eye disease, whether the diagnosis is known or not, to determine if they are eligible for other NEI research studies. No treatment is offered in this study.

People of all ages with various eye conditions, including genetic conditions, eye movement disorders, inflammatory eye diseases, retinal diseases and external eye diseases, may be eligible for this study.

Participants undergo various tests and procedures to diagnose or evaluate their eye disease. The procedures may include the following:

* Personal and family medical history
* Physical examination and blood tests, including genetic testing.
* Eye examination with dilation to measure visual acuity and eye pressure and to examine the front and back parts of the eye.
* Questionnaire about vision and daily activities.
* Conjunctival swab or lacrimal bland biopsy, or both: A sample of cells from the eyes is collected by swabbing the surface of the eye or by surgically removing a small sample of the surface of the eye or tear gland.
* Electroretinogram to examine retinal function: The subject sits in the dark with his or her eyes patched for 30 minutes. The patches are removed, the surface of the eyes is numbed, and contact lenses that can sense signals from the retina are placed on the eyes. The subject then watches flashing lights.
* Fluorescein angiography to examine the blood vessels in the eye: A dye is injected into a vein in the arm. The dye travels through the veins to the blood vessels in the eyes. A camera takes pictures of the dye as it flows through the blood vessels.
* Optical coherence tomography to measure retinal thickness: A machine used to examine the eyes produces cross-sectional pictures of the retina.
* Microperimetry to test how sensitive different parts of the retina are to changing levels of light. The subject sits in front of a computer and presses a button when he or she sees a light on the screen.
* Oculography to record eye movements: Eye movements are measured by contact lenses or goggles that the subject wears while watching a series of spots on a computer screen.

DETAILED DESCRIPTION:
This protocol is designed for the screening of potential research participants with or without a defined diagnosis. This protocol will serve as a point of entry for individuals who may be eligible and wish to participate in the National Eye Institute (NEI) clinical research studies.

Patients who are referred or self-referred will be screened and evaluated during the screening process to determine whether they are suitable participants for any of the ongoing NEI research studies. The screening process may include past and current medical history, a physical examination, diagnostic procedures, and required testing used to establish a patient s diagnosis and determine his/her potential eligibility for research participation. Once the screening process is complete, patients will be informed of their options to participate in one or more of the NEI's current clinical research protocols or natural history studies. If no appropriate research protocol is available for their participation, the patient may receive potential treatment recommendations, which will be shared with the patient s primary provider and referring physician.

This protocol's secondary aim is to collect and store human biospecimens and health information for basic science laboratory research and to generate and test hypotheses. Through such studies, research investigators hope to find possible new ways to detect, treat, and even prevent or cure ophthalmological diseases. Genetic and genomic testing, and biospecimen samples such as blood, body fluid (e.g., urine), and tissue (e.g., skin) may be collected from affected or unaffected adult participants. Biospecimen samples can be obtained at the time of screening or any time after screening. These samples, combined with other clinical data, may be used for basic science laboratory research or stored and used in future research studies. Biospecimen sample collection is voluntary for all participants.

ELIGIBILITY:
* INCLUSION CRITERIA:

Participants will be able to enroll if they:

* Have a diagnosed ocular disease/disorder; OR
* Potentially have an unusual, interesting, or unknown ocular condition that requires the establishment of a diagnosis; OR
* Potentially participate as a disease-free control participant in an NEI clinical research study; OR
* Are an unaffected first-degree relative of a participant with either a diagnosed or undiagnosed ocular disorder; AND
* Have the ability to understand and sign an informed consent OR if they are minor children have a legal parent/guardian with the ability to do the same.
* Adults with impaired capacity to consent must have a Legally Authorized Representative (LAR) who is able to provide informed consent.

EXCLUSION CRITERIA:

Participants will be unable to enroll if they:

* Are unwilling or unable to cooperate with the study procedures.
* Female participants of childbearing potential who are pregnant are not eligible for enrollment.

Ages: 2 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participants can be self-referred or be referrals from medical practitioners, clinics, hospitals, or medical institutions.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2008-08-20 (Actual)

PRIMARY OUTCOMES:
ascertain eligibility | At screening
  Determine eligibility for additional NEI protocols.

CONTACTS AND LOCATIONS:
Overall Officials: Awilda V Holland, R.N., Principal Investigator — National Eye Institute (NEI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2008-EI-0102.html